CLINICAL TRIAL: NCT03426540
Title: Safety and Efficacy of Intravitreal Conbercept Injection After Vitrectomy for the Treatment of Early Proliferative Diabetic Retinopathy
Brief Title: Intravitreal Conbercept After Vitrectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Zhenchuan Zheng, Tianjin Medical University Eye Hospital, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016KY-09
Record Dates: First submitted 2018-01-26; First posted 2018-02-08 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Early Proliferative Diabetic Retinopathy
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conbercept (Experimental): intravitreal conbercept (10 mg/mL, 0.5 mg) immediately after surgery
  Interventions: Drug: Conbercept
- control group (No Intervention): Pars plana vitrectomy alone

INTERVENTIONS:
Drug: Conbercept — Three-port 25-G PPV was performed in all patients using a Constellation system. Patients in the treatment group received an intravitreal injection of conbercept (10 mg/mL, 0.5 mg) using a sterile technique after 25-G vitrectomy.
  Arms: Conbercept

SUMMARY:
To evaluate the safety and efficacy of intravitreal conbercept after vitrectomy for the management of early-stage proliferative diabetic retinopathy (PDR).

Hypothesis: intravitreal conbercept therapy may promote functional and anatomic recovery from PDR. intravitreal conbercept therapy may be a useful and safe method for improving visual outcomes of surgery for early-stage PDR.

DETAILED DESCRIPTION:
The drug conbercept (an anti-vascular endothelial growth factors) was recently made available for management of early prolific diabetic retinopathy, but its safety and efficacy still require study. Therefore, the aim is to evaluate the safety and efficacy of intravitreal conbercept after vitrectomy for the management of early proliferative diabetic retinopathy.The patients were randomly assigned (25 eyes each group) to either treatment group and control after they provided informed consent. The treatment group received intravitreal conbercept (10 mg/mL, 0.5 mg) immediately after surgery, while the control group did not.

At the time of study enrollment, physical examinations, best-corrected visual acuity (BCVA), intraocular pressure and central retinal thickness will be measured and fundoscopy be performed.

The patients are going to be followed up for at least 6 months via BCVA measurement, fundoscopy, OCT, physical examinations and postoperative complications

ELIGIBILITY:
Inclusion Criteria:

1. We enrolled 50 eyes from 50 patients that were affected by VH as a consequence of early active PDR.
2. Patients with non-clearing VH and fibrocellular proliferation without TRD who underwent PPV at Tianjin Medical University Eye Hospital were included in the study.

Exclusion Criteria:

1. A history of previous PPV;
2. Severe intraoperative complications
3. Postoperative silicone oil tamponade;
4. Menstruation;
5. Stroke, a thromboembolic event, or myocardial infarction in the previous
6. months contraindicating the withdrawal of anti-platelet and anti-coagulant medications.

Ages: 28 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
best corrected visual acuity | baseline to 24 weeks post-surgery
  BCVA using a Landolt C acuity chart method

SECONDARY OUTCOMES:
postoperative complications | baseline to 24 weeks post-surgery
  postoperative complications
central retinal thickness | baseline to 24 weeks post-surgery
  Optical coherence tomography (OCT) is an established medical imaging technique that uses light to capture micrometer-resolution, one-dimensional images

CONTACTS AND LOCATIONS:
Overall Officials: Rong X Li, MD,PhD, Principal Investigator — Tianjin Medical University

IPD SHARING:
Plan to Share IPD: No